CLINICAL TRIAL: NCT04580108
Title: Highly Sensitive Serum Cardiac Troponin T and Cardiovascular Events in Patients With Systemic Lupus Erythematosus
Acronym: TROPOPLUS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: NI17026J
Record Dates: First submitted 2020-05-19; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Cardiovascular risk; Biomarkers; Troponin T
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with systemic lupus erythematosus: Patients with systemic lupus erythematosus enrolled in the PLUS cohort between 2007 and 2010

SUMMARY:
Identification of biological markers able to better stratify cardiovascular risks in systemic lupus erythematosus patients is needed. We aimed to determine whether serum cardiac troponin T levels measured with a highly sensitive assay (HS-cTnT) may predict cardiovascular events in systemic lupus erythematosus.

DETAILED DESCRIPTION:
Cardiac Troponin (cTnT) is a marker of myocyte necrosis and injury in the early phase of acute myocardial infarction. Measured with high-sensitivity (HS) assays, HS-cTnT has proven predictive value for coronary heart disease, heart failure, and mortality in the general population at apparent low-risk for cardiovascular events. In a previous study, our group showed that HS-cTnT concentration was associated with subclinical atherosclerosis in systemic lupus erythematosus patients. The aim of this study was to determine whether HS-cTnT was associated with incident cardiovascular events in systemic lupus erythematosus

ELIGIBILITY:
Inclusion Criteria:

* Patient with a systemic lupus erythematosus

Exclusion Criteria:

* Inadequate follow-up period (< 20 months) -past history of CVE at baseline for inclusion in the TROPOPLUS study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with systemic lupus erythematosus
Sampling Method: Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2007-07-03 (Actual); Primary Completion 2012-01-17 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the occurrence of cardiovascular events over follow-up. | Up to 10 years
  Incidents cardiovascular events (CVE) were ascertained by physician interview using a standardized questionnaire and through examination of medical records. cardiovascular events included coronary heart disease, stroke, revascularization procedure for other atherosclerotic cardiovascular diseases and sudden cardiac death. Coronary heart disease was defined as a history of angina, coronary revascularization, or myocardial infarction. All CVE that occurred through March 2019 were considered for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Karim Sacré, MD, PhD, Principal Investigator — GH Bichat-Claude Bernard, Paris, France, 75018
Locations (1):
- Bichat Hospital, Paris, France